CLINICAL TRIAL: NCT06495151
Title: Evaluation of Serum and Peritoneal Fluid Mannose-binding Lectin Associated Serine Protease-3, Adipsin, Properdin, and Complement Factor H Levels in Endometriosis Patients
Brief Title: Endometriosis and Complement System
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Merve Didem Eşkin Tanrıverdi, Medical Doctor, Ankara City Hospital Bilkent
Other Study IDs: E2-22-1998
Record Dates: First submitted 2024-07-03; First posted 2024-07-10 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Endometriosis; Complement System; Alternative Complement Pathway
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples were collected via antecubital venous blood sampling. In the study group, serum samples were obtained just before laparoscopy, while peritoneal fluid (PF) samples were collected from the Douglas pouch at the time of trochar insertion into the abdominal cavity. Serum and PF MASP-3, adipsin, properdin, and CFH levels were evaluated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endometriosis group (Study group): * The study group included 32 women with endometriosis.
  * The study group consisted of women diagnosed with endometriosis who consecutively underwent laparoscopic endometriosis surgery.
  Interventions: Diagnostic Test: Mannose-binding lectin-associated serine protease-3 (MASP-3) Level; Diagnostic Test: Adipsin Level; Diagnostic Test: Properdin Level; Diagnostic Test: Complement Factor H (CFH) Level; Diagnostic Test: Cancer Antigen 125 (CA-125) Level
- Healthy women (Control group): * Control group consisted of 26 healthy women.
  * The control group consisted of women who consecutively visited the outpatient clinic for routine gynecologic examinations and had no known diseases.
  Interventions: Diagnostic Test: Mannose-binding lectin-associated serine protease-3 (MASP-3) Level; Diagnostic Test: Adipsin Level; Diagnostic Test: Properdin Level; Diagnostic Test: Complement Factor H (CFH) Level; Diagnostic Test: Cancer Antigen 125 (CA-125) Level

INTERVENTIONS:
Diagnostic Test: Mannose-binding lectin-associated serine protease-3 (MASP-3) Level — Measurement of venous blood serum and peritoneal fluid levels of MASP-3 level by ELISA method.
Diagnostic Test: Adipsin Level — Measurement of venous blood serum and peritoneal fluid levels of adipsin level by ELISA method.
Diagnostic Test: Properdin Level — Measurement of venous blood serum and peritoneal fluid levels of properdin level by ELISA method.
Diagnostic Test: Complement Factor H (CFH) Level — Measurement of venous blood serum and peritoneal fluid levels of CFH level by ELISA method.
Diagnostic Test: Cancer Antigen 125 (CA-125) Level — Measurement of venous blood serum level of CA-125 level by ELISA method.

SUMMARY:
Endometriosis is a chronic gynecological condition affecting nearly 10% of women of reproductive age. A definitive diagnosis of endometriosis requires laparoscopy. Studies aim to identify novel biomarkers to aid in the development of effective noninvasive diagnostic methods. Despite several theories, the full understanding of the etiopathogenesis remains elusive. A distorted immune response is thought to play a crucial role in the pathophysiology of endometriosis. This study aimed to evaluate whether the levels of alternative complement molecules change in the blood serum and peritoneal fluid of endometriosis patients compared to healthy subjects.

DETAILED DESCRIPTION:
Endometriosis is a chronic gynecological condition affecting nearly 10% of women of reproductive age. It has been reported to contribute to 21-47% of cases of female infertility and 71-87% of cases involving chronic pelvic pain. The definitive diagnosis of endometriosis requires laparoscopy. While CA-125 has diagnostic value, it is not specific to endometriosis. Therefore, studies are focused on identifying novel biomarkers to aid in the development of effective noninvasive diagnostic methods. Despite numerous theories, the etiopathogenesis of endometriosis remains incompletely understood. A distorted immune response is believed to play a crucial role in the pathophysiology of the condition. Regarding alterations in the classical and lectin-dependent complement systems, C3a, C3c, C4, and C5b-9 have been suggested to hold potential diagnostic value in endometriosis. Alternative pathway is another way for complement activation. This study aimed to investigate whether there are alterations in the levels of alternative complement molecules in both the blood serum and peritoneal fluid of patients diagnosed with endometriosis, comparing these levels to those found in healthy individuals. The research focused on understanding potential differences that could contribute to the pathophysiology of endometriosis, aiming to provide insights into the role of the alternative complement pathway in this gynecological condition.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of endometriosis for study group who underwent laparoscopic endometriosis surgery
* Healthy women for control group

Exclusion Criteria:

* Cardiovascular diseases including hypertension
* Type 1 or type 2 diabetes mellitus
* Morbid obesity
* Primary adrenal insufficiency
* Uterine fibroids
* Thyroid dysfunctions including Hashimoto thyroiditis and Grave's disease
* Hepatic dysfunctions
* Renal insufficiency
* Genetic disorders in chromosome constitution or karyotype analysis including monosomy X, trisomy X and gene mutations as BMP15, FMR I, POFIB, and GDF9
* Neurologic diseases
* Psychiatric disorders
* Autoimmune diseases or syndromes including Addison's disease, autoimmune syndromes, scleroderma, Sjogren's syndrome, myasthenia gravis, inflammatory bowel diseases, multiple sclerosis, rheumatoid arthritis, systemic lupus erythematosus and familial Mediterranean fever
* History of any malignancy
* History of exposure to chemotherapeutic agents or radiotherapy

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Endometriosis is the presence of endometrial tissue outside the uterus, such as in the ovaries, fallopian tubes, peritoneal membrane, or abdominal cavity, and it is diagnosed exclusively in females.
Study Population: Study population includes a total of 58 participants. The study group consists of 32 women with the diagnosis of endometriosis, and the control group consists of 26 healthy women.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2022-10-07 (Actual)

PRIMARY OUTCOMES:
Serum and peritoneal fluid mannose-binding lectin-associated serine protease-3 level | day 1
  Nanogram/milliliter
Serum and peritoneal fluid adipsin level | day 1
  Nanogram/milliliter
Serum and peritoneal fluid properdin level | day 1
  Nanogram/milliliter
Serum and peritoneal fluid complement factor H level | day 1
  Nanogram/milliliter

SECONDARY OUTCOMES:
Serum cancer antigen 125 level | day 1
  Unit/milliliter

CONTACTS AND LOCATIONS:
Overall Officials: Merve Didem Eşkin Tanrıverdi, MD, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD are available which may be shared in necessary conditions.

REFERENCES:
- [Background] Falcone T, Flyckt R. Clinical Management of Endometriosis. Obstet Gynecol. 2018 Mar;131(3):557-571. doi: 10.1097/AOG.0000000000002469. PMID 29420391
- [Background] Chapron C, Marcellin L, Borghese B, Santulli P. Rethinking mechanisms, diagnosis and management of endometriosis. Nat Rev Endocrinol. 2019 Nov;15(11):666-682. doi: 10.1038/s41574-019-0245-z. Epub 2019 Sep 5. PMID 31488888
- [Background] Karadadas E, Hortu I, Ak H, Ergenoglu AM, Karadadas N, Aydin HH. Evaluation of complement system proteins C3a, C5a and C6 in patients of endometriosis. Clin Biochem. 2020 Jul;81:15-19. doi: 10.1016/j.clinbiochem.2020.04.005. Epub 2020 Apr 20. PMID 32325082
- [Background] Kabut J, Kondera-Anasz Z, Sikora J, Mielczarek-Palacz A. Levels of complement components iC3b, C3c, C4, and SC5b-9 in peritoneal fluid and serum of infertile women with endometriosis. Fertil Steril. 2007 Nov;88(5):1298-303. doi: 10.1016/j.fertnstert.2006.12.061. Epub 2007 May 4. PMID 17482181
- [Background] Xu Y, Ma M, Ippolito GC, Schroeder HW Jr, Carroll MC, Volanakis JE. Complement activation in factor D-deficient mice. Proc Natl Acad Sci U S A. 2001 Dec 4;98(25):14577-82. doi: 10.1073/pnas.261428398. Epub 2001 Nov 27. PMID 11724962
- [Background] Ricklin D, Hajishengallis G, Yang K, Lambris JD. Complement: a key system for immune surveillance and homeostasis. Nat Immunol. 2010 Sep;11(9):785-97. doi: 10.1038/ni.1923. Epub 2010 Aug 19. PMID 20720586
- [Background] Poppelaars F, Faria B, Schwaeble W, Daha MR. The Contribution of Complement to the Pathogenesis of IgA Nephropathy: Are Complement-Targeted Therapies Moving from Rare Disorders to More Common Diseases? J Clin Med. 2021 Oct 14;10(20):4715. doi: 10.3390/jcm10204715. PMID 34682837
- [Background] Liu M, Luo X, Xu Q, Yu H, Gao L, Zhou R, Wang T. Adipsin of the Alternative Complement Pathway Is a Potential Predictor for Preeclampsia in Early Pregnancy. Front Immunol. 2021 Oct 4;12:702385. doi: 10.3389/fimmu.2021.702385. eCollection 2021. PMID 34671343
- [Background] Gursoy Calan O, Calan M, Yesil Senses P, Unal Kocabas G, Ozden E, Sari KR, Kocar M, Imamoglu C, Senses YM, Bozkaya G, Bilgir O. Increased adipsin is associated with carotid intima media thickness and metabolic disturbances in polycystic ovary syndrome. Clin Endocrinol (Oxf). 2016 Dec;85(6):910-917. doi: 10.1111/cen.13157. Epub 2016 Aug 15. PMID 27434652
- [Background] Zhang J, Teng F, Pan L, Guo D, Liu J, Li K, Yuan Y, Li W, Zhang H. Circulating adipsin is associated with asymptomatic carotid atherosclerosis in obese adults. BMC Cardiovasc Disord. 2021 Oct 25;21(1):517. doi: 10.1186/s12872-021-02329-3. PMID 34696714
- [Background] Barratt J, Weitz I. Complement Factor D as a Strategic Target for Regulating the Alternative Complement Pathway. Front Immunol. 2021 Sep 9;12:712572. doi: 10.3389/fimmu.2021.712572. eCollection 2021. PMID 34566967
- [Background] Lei X, Song X, Fan Y, Chen Z, Zhang L. The Role and Potential Mechanism of Complement Factor D in Fibromyalgia Development. J Pain Res. 2023 Dec 19;16:4337-4351. doi: 10.2147/JPR.S439689. eCollection 2023. PMID 38145036
- [Background] Agostinis C, Balduit A, Mangogna A, Zito G, Romano F, Ricci G, Kishore U, Bulla R. Immunological Basis of the Endometriosis: The Complement System as a Potential Therapeutic Target. Front Immunol. 2021 Jan 11;11:599117. doi: 10.3389/fimmu.2020.599117. eCollection 2020. PMID 33505394
- [Background] Chen LH, Lo WC, Huang HY, Wu HM. A Lifelong Impact on Endometriosis: Pathophysiology and Pharmacological Treatment. Int J Mol Sci. 2023 Apr 19;24(8):7503. doi: 10.3390/ijms24087503. PMID 37108664
- [Background] Garred P, Genster N, Pilely K, Bayarri-Olmos R, Rosbjerg A, Ma YJ, Skjoedt MO. A journey through the lectin pathway of complement-MBL and beyond. Immunol Rev. 2016 Nov;274(1):74-97. doi: 10.1111/imr.12468. PMID 27782323